CLINICAL TRIAL: NCT01489488
Title: Relative Bioavailability and Food Effect Study of Two Oral Liquid Formulations in Comparison to a 1 mg Tablet of Riociguat to Characterize Its Pharmacokinetic Properties in Healthy Male and Female Adult Subjects in a Randomized, Open Label, 5-fold Crossover Design
Brief Title: Relative Bioavailability and Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 14986; 2011-001893-24 (EudraCT Number)
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Pharmacology, Clinical
Keywords: Relative bioavailability study
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)
- Arm 2 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)
- Arm 3 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)
- Arm 4 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)
- Arm 5 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (BAY63-2521) — Single oral dose of 2.4 milligram (mg) riociguat (BAY63-2521) as pediatric high-concentration suspension (0.15 mg per milliliter [mg/mL], i.e. 16 mL) under fasting conditions
  Arms: Arm 1
Drug: Riociguat (BAY63-2521) — Single oral dose of 2.4 mg riociguat as pediatric high-concentration suspension (0.15 mg/mL, i.e. 16 mL) under fed conditions
  Arms: Arm 2
Drug: Riociguat (BAY63-2521) — Single oral dose of 0.3 mg riociguat as pediatric high-concentration suspension (0.15 mg/mL, i.e. 2 mL) under fasting conditions
  Arms: Arm 3
Drug: Riociguat (BAY63-2521) — Single oral dose of 0.15 mg riociguat as pediatric low-concentration suspension (0.03 mg/mL, i.e. 5 mL) under fasting conditions
  Arms: Arm 4
Drug: Riociguat (BAY63-2521) — Single oral dose of riociguat immediate release (IR) tablet 1 mg under fasting conditions
  Arms: Arm 5

SUMMARY:
Primary objective: To determine oral bioavailability of the liquid formulation intended for pediatric use and potential food effects in healthy adults.

Secondary objective: To evaluate safety and tolerability measured by physical examination findings, vital signs, electrocardiogram (ECG), laboratory parameters, and adverse events (AEs).

DETAILED DESCRIPTION:
Clinical pharmacology

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers
* Age 18-45 years
* Body mass index (BMI) 18.0-29.9 kg/m²
* Systolic blood pressure (SBP) 110-145 mmHg
* No drugs 2 weeks before treatment
* Nonsmokers for at least 12 weeks

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Medical disorder that would impair the subject's ability to complete the study in the opinion of the Investigator
* Known hypersensitivity to the study drugs (active substance or excipients of the preparations)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Relevant diseases within the last 4 weeks prior to the first study drug administration
* Regular use of medicines
* Regular use of therapeutic or recreational drugs
* Use of any medication within the 2 weeks preceding the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC) of Riociguat and its Analyte M1 (BAY60-4552) | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC is defined as area under concentration versus time curve from time 0 (predose) to extrapolated infinite time. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration (Cmax) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of plasma samples and measuring the concentrations of drug in each sample. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Infinity Divided by Dose (AUC/D) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration Adjusted by Dose (Cmax/D) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Zero to Infinity Divided by Dose per Kilogram Body Weight (AUC,norm) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  AUC is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption. AUCnorm is defined as AUC divided by dose per kg body weight.
Maximum Observed Plasma Concentration Divided by Dose per Kilogram Body Weight (Cmax,norm) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Cmax,norm is defined as Cmax divided by dose per kg body weight.
Time to Reach Maximum Drug Concentration in Plasma (tmax) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Terminal Half Life (t1/2) of Riociguat and its Analyte M1 (BAY60-4552) | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  Half life associated with terminal slope refers to the elimination of the drug. It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase of elimination. It is expressed in hours and derived from the terminal slope of the concentration versus time curve. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Mean Residence Time (MRT) of Riociguat and its Analyte M1 (BAY604552) | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  MRT is an average duration of the drug in the body, and is expressed in hours.
Area Under the Concentration Versus Time Curve From Zero to Last Quantifiable Concentration (AUC[0-tlast]) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-tlast) is defined as AUC from time zero to the last data point above the lower limit of quantification. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Last Quantifiable Concentration Divided by Dose per Kilogram Body Weight (AUC[0-tlast]norm) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-tlast), norm is defined as AUC from time zero to the last data point above the lower limit of quantification divided by dose per kg body weight. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Last Quantifiable Concentration Divided by Dose (AUC[0-tlast]/D) of Riociguat and its Analyte M1 (BAY60-4552) After a Single Dose | 0 hour (predose), 15, 30, 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 12, 15, 24, 36, 48, and 72 hours postdose
  AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-tlast)/D is defined as AUC from time zero to the last data point above the lower limit of quantification divided by dose. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/